CLINICAL TRIAL: NCT03483389
Title: Immune Activation and Neurodegeneration in HIV Infection and Heavy Drinking
Brief Title: Alcohol and Immune Response
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brown University (Other)
Responsible Party: Principal Investigator, Mollie Monnig, Assistant Professor of Behavioral and Social Sciences, Brown University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: 1710001919
Record Dates: First submitted 2018-03-06; First posted 2018-03-30 (Actual); Last update posted 2021-07-27 (Actual); Status verified 2021-07

CONDITIONS: Alcohol Drinking; Alcohol; Harmful Use
MeSH Terms: conditions — Alcohol Drinking | interventions — Ethanol

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Alcohol, placebo (Experimental): Alcohol, ethyl - Placebo
  Interventions: Drug: Alcohol, Ethyl; Other: Alcohol, Ethyl - placebo
- Alcohol, low dose (Experimental): Alcohol, ethyl - Low dose
  Interventions: Drug: Alcohol, Ethyl; Other: Alcohol, Ethyl - placebo
- Alcohol, moderate dose (Experimental): Alcohol, ethyl - Moderate dose
  Interventions: Drug: Alcohol, Ethyl; Other: Alcohol, Ethyl - placebo

INTERVENTIONS:
Drug: Alcohol, Ethyl — Randomized within-subjects design
  Other Names: Alcohol
Other: Alcohol, Ethyl - placebo — Randomized within-subjects design
  Other Names: Placebo

SUMMARY:
This study investigates how alcohol affects the immune system and behavior in healthy adults. The study also will examine how an individual's typical drinking habits may affect the immune system's response to alcohol.

ELIGIBILITY:
Inclusion Criteria:

* Ages 21-55 years
* Able to speak and read English
* Regular use of alcohol
* Weight > or = to 110 lbs and body mass index (BMI) in the 18.5-30 kg/m2 range
* No self-reported use of drugs

Exclusion Criteria:

* Currently seeking treatment for alcohol or drug use
* Chronic disease
* Use of certain medications
* GI disorders
* Daily/near-daily use of NSAIDs
* Positive urine test for certain drugs
* History of withdrawal symptoms precipitated by alcohol abstinence
* Clinical Institute Withdrawal Assessment for Alcohol score greater than or equal to 10
* History of seizures
* Current major psychiatric disorder
* History of adverse reaction to standard blood draw
* Inability to abstain from tobacco for 8 hours
* Inability to abstain from cannabis for 48 hours
* Pregnant, breastfeeding, or may become pregnant

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 76 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2021-06-18 (Actual); Study Completion 2021-06-18 (Actual)

PRIMARY OUTCOMES:
Plasma lipopolysaccharide (pg/ml) | 0-4 hours
  Plasma concentration of lipopolysaccharide, measured in picograms/ml
Plasma lipopolysaccharide binding protein (ng/ml) | 0-4 hours
  Plasma concentration of lipopolysaccharide binding protein, measured in nanograms/ml
Soluble cluster of differentiation 14 (ng/ml) | 0-4 hours
  Plasma concentration of soluble cluster of differentiation 14, measured in nanograms/ml
Soluble cluster of differentiation 163 (ng/ml) | 0-4 hours
  Plasma concentration of soluble cluster of differentiation 163, measured in nanograms/ml

SECONDARY OUTCOMES:
Response time in ms | 0-4 hours
  Response time in milliseconds, as measured by the NIH Toolbox and Cued Go/No-Go test

CONTACTS AND LOCATIONS:
Locations (1):
- Brown University, Providence, Rhode Island, United States